CLINICAL TRIAL: NCT03391323
Title: Medacta GMK Sphere® Medial-Pivot, Cruciate Substituting vs. Medacta GMK PS Posterior Stabilized Kne vs. OMNI Apex Knee Ultracongruent vs. Triathlon® Posterior Stabilized & Cruciate Substituting Outcomes Study
Brief Title: Medacta GMK Sphere® vs. Medacta GMK PS Post-Market Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David F. Scott, MD (Other)
Collaborators: Medacta USA (Industry)
Responsible Party: Sponsor-Investigator, David F. Scott, MD, Principal Investigator, Spokane Joint Replacement Center
Organization: Spokane Joint Replacement Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SJRC-GMK
Record Dates: First submitted 2017-12-11; First posted 2018-01-05 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Joint Disease
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Medacta GMK Sphere® Medial-Pivot Knee Prosthesis (Other)
  Interventions: Device: Medacta GMK Sphere® Medial-Pivot Knee Prosthesis
- Medacta GMK PS Posterior Stabilized Knee Prosthesis (Other)
  Interventions: Device: Medacta GMK PS Posterior Stabilized Knee Prosthesis

INTERVENTIONS:
Device: Medacta GMK Sphere® Medial-Pivot Knee Prosthesis
  Arms: Medacta GMK Sphere® Medial-Pivot Knee Prosthesis
Device: Medacta GMK PS Posterior Stabilized Knee Prosthesis
  Arms: Medacta GMK PS Posterior Stabilized Knee Prosthesis

SUMMARY:
The study is a prospective, randomized comparison of total knee arthroplasty with the Medacta GMK Sphere® knee compared to the Medacta GMK PS knee, with comparison to data from previous trials of similar study design.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the Informed Consent.
* Patients able to comply with follow-up requirements including postoperative weight bearing restrictions and self-evaluations.
* Male and non-pregnant female patients ages 21 - 80 years of age at the time of surgery.
* Patients requiring a primary total knee replacement.
* Patients with a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
* Patients with intact collateral ligaments.

Exclusion Criteria:

* Patients with inflammatory arthritis.
* Patients that are morbidly obese, body mass index (BMI) > 40.
* Patients with a history of total or unicompartmental reconstruction of the affected joint.
* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
* Patients that are immunologically compromised, or receiving chronic steroids (>30 days), excluding inhalers.
* Patients bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prosthesis.
* Patients with knee fusion to the affected joint.
* Patients with an active or suspected latent infection in or about the knee joint.
* Patients whose surgery will utilize computer-assisted surgical navigation (CAOS) techniques.
* Patients whose surgery will utilize minimally invasive surgical techniques.
* Patients that are prisoners.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Forgotten Joint Score (FJS) | Change from baseline at 2 years and 5 years post-operative
  The average Forgotten Joint Score (FJS) of those patients receiving the Medacta GMK Sphere® knee prosthesis will be compared with the average FJS of those receiving the Medacta GMK PS knee prosthesis.
  The FJS total score range is 0-100, with higher scores indicating a higher degree of "forgetting" the artificial joint, that is, a lower degree of awareness.

SECONDARY OUTCOMES:
Total Knee Society Score (KSS) | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Clinical outcomes will be evaluated via the Knee Society Score (KSS). The KSS is subdivided into a Knee Assessment score which rates only the knee joint itself, and a Functional Assessment score which rates the subject's ability to walk and climb stairs. Both scores range from 0-100, with a higher score indicating a better outcome.
Lower Extremity Activity Scale (LEAS) | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Clinical outcomes will be evaluated via the Lower Extremity Activity Scale (LEAS). The LEAS scale range is 1-18, with a higher value indicating a higher level of activity.
Radiographic Analysis | Pre-operative, 6 weeks, 6 months, 1, 2, 3, 4, and 5 years post-operative
  Radiographs will be assessed for radiolucency, migration and subsidence. An AP Longstanding view will be obtained pre-operatively, and at 6 weeks and 1 year post-operatively to determine degree of Varus or Valgus.

CONTACTS AND LOCATIONS:
Overall Officials: David Scott, MD, Principal Investigator — Spokane Joint Replacement Center
Locations (1):
- Spokane Joint Replacement Center, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No